CLINICAL TRIAL: NCT03273959
Title: Effects Of An Exercise Program During The Hospitalization Of Children And Adolescents With Cystic Fibrosis: Randomized Clinical Test
Brief Title: Program Of Exercises During The Hospitalization Of Children And Adolescents With Cystic Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0126
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis in Children; Cystic Fibrosis Pulmonary Exacerbation; Cystic Fibrosis With Exacerbation
Keywords: Physiotherapy; Physical Therapy; Exercise; Hospitalization; Pediatric; Adolescents
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups: control and intervention.
Who Masked: Investigator
Masking Description: The evaluator who will apply the tests at the beginning and end of the hospital stay will be blinded. The evaluator who will apply the tests at the beginning and end of the hospital stay will be blinded. Another health professional who will participate in the research will apply the protocol of supervised exercises in patients who are randomized to the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group control (No Intervention): Patients randomized to the control group will receive routine physiotherapeutic follow-up, performed by the physiotherapist of the hospital during the hospitalization period. Supervision includes inhalation therapy and respiratory physiotherapy. Respiratory exercises and thoracic maneuvers for bronchial hygiene will be performed, according to what the patient is accustomed to perform. Other techniques besides these can be added at the discretion of the physiotherapist according to the needs of the patient. In pediatric hospitalization patients also receive care from physical educators who associate recreational and recreational activities with the treatment.
- Intervention group (Experimental): Patients randomized to the intervention group, in addition to routine physical therapy follow-up, will receive a program of physical exercises, illustrated in the form of a booklet and guided by a health professional. The patient is instructed to perform physical exercises five times a week until a hospital discharge. The participant will receive with a booklet a diary to write down the days in which to carry out the proposed exercises, in case of fault he will write down the reason for not performing. The exercise protocol includes: Punching, climbing and descending steps, sit and stand, push-ups on the wall, stationary gait, abdominal, physiotherapy bridge, jumping on the floor ladder, cycling on the cycle ergometer and stretching.
  Interventions: Other: Exercise protocol

INTERVENTIONS:
Other: Exercise protocol — Protocol of exercises performed in hospital admission in children and adolescents with cystic fibrosis in the exacerbation phase.
  Arms: Intervention group

SUMMARY:
The objective of this study was to evaluate the effect of a physical exercise program on the functional capacity of children and adolescents with cystic fibrosis hospitalized at the Hospital de Clínicas of Porto Alegre (HCPA) through a six-minute walk test using the distance traveled In six minutes.

In the first 48 hours of hospital stay, the following evaluations will be performed: Six-minute walk test, physical and health fitness test, spirometry and data collection. Patients will be randomized to either control group or intervention group. The control group will receive the conventional treatment offered by hospital care, the intervention group will receive this same treatment plus an exercise protocol. After 14 days they will be reevaluated with the same tests applied at the beginning of hospitalization.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the effect of a protocol of physical exercises on the functional capacity of children and adolescents with cystic fibrosis, hospitalized, in the stage of exacerbation of the disease.

In the first 48 hours of hospitalization patients and their caregivers will be invited to participate in the study. We will start with the following evaluations: Six-minute walk test, spirometry, physical fitness and health test (includes: walking, abdominal, flexibility and abdominal circumference), clinical score of shwachman kulczycki and Collected data from medical records.

After the initial evaluation the patient will be randomized to control group or intervention group. The control group will receive the conventional physiotherapy by the assistance team and the recreation service by the physical education. The intervention group will receive the same assistance plus the intervention with the exercise protocol five times a week supervised by a health professional. The exercise protocol includes: Punching, climbing and descending steps, sit and stand, push-ups on the wall, stationary gait, abdominal, physiotherapy bridge, jumping on the floor ladder, cycling on the cycle ergometer and stretching.

At hospital discharge both groups will repeat the initial tests. The hypothesis is that the intervention group showed an improvement in functional capacity compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* They will be included in the study of patients from 6 to 18 years old, regularly followed by the Pediatric Pulmonology team of the HCPA, with diagnosis of cystic fibrosis according to the consensus criteria admitted to hospital admission due to exacerbation of the disease.
* Hospital admission is defined as a stay of 24 hours or more in any HCPA unit.
* An exacerbation of lung disease is defined as the presence of one or more of the following: Change in sputum volume and color, new or enlarged hemoptysis, increased cough, increased dyspnoea, malaise, fatigue, lethargy, fever, anorexia or Loss of weight, headache or pain in the sinuses, alteration of the pulmonary auscultation, non-FEV1 decrease of more than 10%, radiological, eradication of new bacteria.

Exclusion Criteria:

* Patients with cardiac, orthopedic or trauma complications that make it impossible to perform the proposed exercises;
* Patients with hemodynamic instability, massive hemoptysis, pneumothorax, and continuous use of noninvasive ventilation.
* Pregnant women

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-08-28 (Estimated); Study Completion 2019-03-28 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | 14 days
  Evaluate the distance covered by the six-minute walk test

SECONDARY OUTCOMES:
Pulmonary functional capacity | 14 days
  Spirometry
Physical fitness and health | 14 days
  Generate a score.
Clinical score Shwachman-Kulczycki | 14 days
  Scoring for general activity, physical examination, nutrition and radiological findings of the thorax.
bacteriology | 14 days
  The last bacteriological exams will be noted
Nutrition assessment | 14 days
  Body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Ziegler, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil